CLINICAL TRIAL: NCT07026318
Title: Endovascular Therapy Combined With Tirofiban for Intracranial Atherosclerotic Acute Ischemic Stroke: A Multicenter, Prospective, Double-blind, Vehicle-controlled, Randomized Controlled Trial
Brief Title: Endovascular Therapy Combined With Tirofiban for Intracranial Atherosclerotic Acute Ischemic Stroke
Acronym: ANGEL-DRUG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANGEL-DRUG
Record Dates: First submitted 2025-06-03; First posted 2025-06-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; Tirofiban; placebo; Randomized Controlled Trial; Intracranial Atherosclerotic
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental): Receive Tirofiban treatment following endovascular therapy
  Interventions: Drug: Tirofiban
- placebo group (Placebo Comparator): Receive placebo treatment after endovascular therapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tirofiban — After endovascular treatment, tirofiban is infused at a rate of 0.4 μg/kg/min for 30 minutes, followed by a maintenance infusion at 0.1 μg/kg/min until 24 hours postoperatively.
  Arms: Tirofiban group
Drug: Placebo — Following endovascular treatment, patients receive normal saline placebo, with the dosage calculated in the same manner as that of tirofiban in the experimental group.
  Arms: placebo group

SUMMARY:
This randomized controlled trial aims to evaluate whether adjunctive tirofiban therapy combined with endovascular treatment (EVT) improves neurological outcomes in patients with acute large vessel occlusion due to large-artery atherosclerosis. Patients will be randomized to receive either tirofiban or matching placebo after EVT. The primary efficacy endpoint is the proportion of patients achieving functional independence (modified Rankin Scale 0-2) at 90±7 days, while the safety endpoint is the probability of symptomatic intracranial hemorrhagewithin 48 hours after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Pre-stroke modified Rankin Scale (mRS) score of 0-1
3. Acute ischemic stroke symptoms present within 24 hours of last known well time
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score ≥6
5. Anterior circulation: Alberta Stroke Program Early CT Score (ASPECTS) ≥6 Posterior circulation: pc-ASPECTS ≥6
6. Occlusion of intracranial internal carotid artery (ICA), M1 segment of middle cerebral artery (MCA), V4 segment of vertebral artery, or basilar artery
7. Clinical care team plans to perform endovascular thrombectomy (EVT)
8. Subject or legally authorized representative can provide informed consent
9. Residual stenosis ≥50% without planned angioplasty/stenting

Exclusion Criteria:

1. Intracranial hemorrhage confirmed by imaging prior to randomization, or major intracranial hemorrhage on intraprocedural flat-panel CT
2. Gastrointestinal or genitourinary bleeding within 30 days post-stroke onset, or major surgery within 14 days
3. Bleeding diathesis including coagulopathy (platelets <100×10⁹/L, aPTT >50s, or INR >2.0), DOAC use within 48 hours, or history of HIT
4. Pregnancy or lactation at admission
5. Contraindications to radiographic contrast agents, nickel, titanium or their alloys
6. Life expectancy <6 months
7. Pre-existing neurological/psychiatric conditions that may confound assessment
8. Severe renal insufficiency (GFR <30mL/min or Scr >220μmol/L [2.5mg/dL])
9. Arterial tortuosity or anomalies preventing device delivery
10. Unlikely to complete 90-day follow-up
11. Any confirmed cardioembolic source (including atrial fibrillation, valvular disease, intracardiac thrombus, recent MI, cardiomyopathy with EF <30%, etc.)
12. Tirofiban or other GP IIb/IIIa inhibitor use before randomization or other GP IIb/IIIa inhibitor used post treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with mRS 0-2 | 90±7 days
  Proportion of patients with Modified Rankin Scale (mRS) 0-2, Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.

SECONDARY OUTCOMES:
Change in NIHSS score from baseline | 36±12 hours post-randomization
  Change in National Institute of Health stroke scale score from baseline.The NIH Stroke Scale (NIHSS) score ranges from 0 to 42 points, with lower scores indicating better neurological function
Vascular recanalization rate assessed by CT/MR angiography | 36±12 hours post-randomization
  Vascular recanalization rate assessed by CT/MR angiography
Change in infarct volume | 7±3 days post-randomization or discharge
  Change in infarct volume
Distribution of mRS scores | 7±3 days/discharge；90±7 days post-randomization
  Modified Rankin Scale（0-6）, A lower MRS score indicates better functional status for the patient.
Proportion of patients achieving mRS 0-1 | 90±7 days
  Proportion of patients achieving mRS 0-1
Proportion of patients achieving mRS 0-3 | 90±7 days
  Proportion of patients achieving mRS 0-3
Incidence of Pharmacologic rescue therapy | 90±7 days
  Incidence of Pharmacologic rescue therapy
Incidence of rescue therapy | 90±7 days
  Incidence of rescue therapy
EQ-5D-5L utility score | 90±7 days
  The EuroQol 5-Dimension 5-Level Utility Score (EQ-5D-5L utility score) ranges from -0.594 to 1.000 (Chinese value set), assessing health-related quality of life, with higher scores indicating better health status.
Probability of symptomatic intracranial hemorrhage | 48 hours
  Probability of symptomatic intracranial hemorrhage (Heidelberg Standards)
All-cause mortality | 90±7 days post-randomization
  All-cause mortality
Probability of any intracranial hemorrhage | 48 hours post-randomization
  Probability of any intracranial hemorrhage (Heidelberg Standards)

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital Affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No